CLINICAL TRIAL: NCT06619275
Title: Ripretinib in Patients With Previously Treated Advanced Gastrointestinal Stromal Tumor (GIST): a Prospective, Longitudinal, Multicenter, Observational Study in Germany
Brief Title: Ripretinib (QINLOCK®) According to Current SmPC
Acronym: INTEREST
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Deciphera Pharmaceuticals (Switzerland) AG (Unknown)
Responsible Party: Sponsor
Other Study IDs: iOM-120455
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: GIST - Gastrointestinal Stromal Tumor
Keywords: advanced
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — ripretinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ripretinib — Switch-Control Tyrosine Kinase Inhibitor

SUMMARY:
The goal of this prospective, observational study INTEREST is to collect real-world data on ripretinib treatment in a broad patient population in Germany. Ripretinib will be administered according to the current SmPC. Thus, INTEREST will evaluate for the first time ripretinib in GIST patients in a real-world setting in Germany.

The main questions the study aims to answer are:

* Evaluate quality of live (QoL) using the questionnaire EQ-5D-5L to gain knowledge about how ripretinib treatment affects GIST patients' well-being (change compared to Baseline, Time to Deterioration)
* Assessment of effectiveness in routine treatment (Progression-Free Survival, Overall Survival, Best Response, Overall Response Rate, Disease Control Rate
* Assessment of drug safety
* Assessment of parameters of physicians' treatment decision making
* Description of treatment reality in detail

ELIGIBILITY:
Inclusion Criteria:

Patient is eligible if all criteria are met:

* Aged 18 years or older.
* Histologically confirmed advanced GIST.
* Patients must have received prior treatment with three or more kinase inhibitors, including imatinib.
* Decision for treatment with ripretinib as per current SmPC.
* Signed written informed consent

  * Patients are allowed to be enrolled up to 6 weeks after their first dose of ripretinib. Patients with signed written informed consent after start of ripretinib treatment are not participating in the PRO assessments.
* Willingness and capability to participate in Patient-Reported Outcome (PRO) assessment in German language.
* Other criteria according to current SmPC.

Exclusion Criteria:

* Participation in an interventional clinical trial within 30 days prior to enrolment or simultaneous participation in an interventional clinical trial except for the follow-up period.
* Patients unable to consent.
* Other contraindications according to current SmPC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with advanced GIST who received 3 or more tyrosine kinase inhibitors (including imatinib).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-08-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Evaluate Quality of Live (QoL): EQ-5D-5L index value | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Evaluation of Quality of Life by validated European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) questionnaire. Change from baseline in the EQ-5D-5L index value
Evaluate Quality of Live (QoL): EQ-Visual Analogue Scale (VAS) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Evaluation of Quality of Life by validated European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) questionnaire. Change from baseline in the EQ-Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
Subjective well-being: EQ-5D-5L questionnaire (index value) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Time to deterioration (TTD) in the EQ-5D-5L index value
Subjective well-being: EQ-5D-5L questionnaire (EQ-VAS) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Time to deterioration (TTD) in the European Quality- Visual Analogue Scale (EQ-VAS)
Assess effectiveness in routine treatment: Progression-free survival (PFS) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  PFS is defined as time interval measured form the day of first ripretinib administration to first progression or death, whichever comes first. Patients without tumor progression or death at the time of analysis will be censored at their date of last contact.
Assess effectiveness in routine treatment: Overall Survival (OS) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  OS is defined as the time interval measured form the day of first ripretinib administration to time of death from any cause. Time to last contact will be used if a patient has no documented date of death and OS for the patient will be considered censored.
Assess effectiveness in routine treatment: Best response | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Best response is defined as Complete Response (CR), Partial Response (PR), Stable Disease (SD), or Progressive Disease (PD))
Assess effectiveness in routine treatment: Overall Response Rate (ORR) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  ORR is defined as the proportion of patients achieving a complete or partial response as best response.
Assess effectiveness in routine treatment: Disease Control Rate (DCR) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  DCR is defined as proportion of patients with Complete Response, Partial Response or Stable Disease as best response.
Assess drug safety: Incidence of (serious) treatment emergent adverse events (TEAEs) | Baseline up to 30 days after ripretinib therapy
  An adverse event will be classified as TEAE if it is related to the study medication (ripretinib).
Assess drug safety: Incidence of (serious) treatment emergent adverse drug reactions (TEADRs) | Baseline up to 30 days after ripretinib therapy
  An adverse drug reaction will be classified as TEADR if it is temporally related to the study medication (ripretinib).
Assess parameters of physicians' treatment decision making using a questionnaire | Baseline
  Frequency of distinct parameters affecting therapy choice; questionnaire completed by treating physician.
Line of ripretinib treatment | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Line of ripretinib treatment
Absolute dose intensity | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Absolute dose intensity of ripretinib
Relative dose intensity | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Relative dose intensity of ripretinib
Frequency of dose modifications | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Frequency of dose modifications during ripretinib treatment
Type of dose modifications | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Type of dose modifications during ripretinib treatment
Reasons of dose modifications | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Reasons of dose modifications during ripretinib treatment
Duration of treatment | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Duration of treatment with ripretinib
Reasons for end of treatment (EOT) | max. 36 months; from the patient-specific study start to end of study (during ripretinib treatment and follow-up)
  Description of treatment reality in detail: Reasons for EOT of treatment with ripretinib
Previous local anticancer therapies per treatment setting | Baseline
  Description of treatment reality in detail: Frequency of previous local anticancer therapies per treatment setting
Previous local anticancer therapies per treatment line | Baseline
  Description of treatment reality in detail: Frequency of previous local anticancer therapies per treatment line
Previous systemic anticancer therapies per treatment setting | Baseline
  Description of treatment reality in detail: Frequency of previous systemic anticancer therapies per treatment setting
Previous systemic anticancer therapies per treatment line | Baseline
  Description of treatment reality in detail: Frequency of previous systemic anticancer therapies per treatment line
Concomitant local anticancer therapies | Baseline up to 30 days after ripretinib therapy
  Description of treatment reality in detail: Frequency of concomitant local anticancer therapies (i.e., surgeries and radiotherapies)
Subsequent local anticancer therapies | From date of end of ripretinib treatment up to 36 months
  Description of treatment reality in detail: Frequency of subsequent local anticancer therapies

CONTACTS AND LOCATIONS:
Locations (1):
- Praxis für interdisziplinäre Onkologie und Hämatologie, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No